CLINICAL TRIAL: NCT00200759
Title: Drug Interactions and Bioavailability of Cranberry
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: R21AT002073-01 (NIH); R21AT002073-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2009-11

CONDITIONS: Healthy; Drug Interactions
Keywords: Vaccinium macrocarpon; Antioxidants; Drug Interactions
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cranberry juice and capsules

SUMMARY:
The purpose of this study is to evaluate the potential of cranberry juice to interact with conventional drugs. This study will also determine the the amount of cranberry flavonoids that appear in the blood and in the urine.

DETAILED DESCRIPTION:
The use of cranberry (CB) juice and powders, both alone and in combination with conventional medicine, has become more common for the treatment of urinary tract infections (UTIs) and and other acute or chronic conditions. Cytochromes P450 enzymes are a group of proteins involved in metabolism of certain substances. A group of cytochrome P-450 (CYP) enzymes are extensively involved in drug metabolism. The pharmacokinetics of many drugs often vary considerably among individuals, largely because of variations in the expression of different cytochrome P-450 (CYP) enzymes in the liver and other tissues. Flavonoids are antioxidants that may have health benefits. The flavonoids may also be responsible for cranberry's effects on urinary tract infections.

To evaluate the drug interaction potential of cranberry, single doses of the three safe probe drugs alprazolam, dextromethorphan, and caffeine will be administered before and after a 14-day treatment period with cranberry powder. Changes in the pharmacokinetics of these probe drugs will indicate the degree of enzyme inhibition or induction. The key pharmacokinetic parameters for four major CB flavonoids will be estimated by following the plasma concentration versus time course of absorbed flavonoids and their excretion in urine. The area under the plasma concentration versus time curve (AUC), oral clearance (Clo), terminal elimination half-life (T1/2) and renal clearance (Clren) will be determined for: epicatechin, quercetin (total glycosides), procyanidin A2, and cyanidin-3-galactoside.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative urine pregnancy test prior to enrollment and must be committed to using barrier methods of birth control throughout the study.

Exclusion Criteria:

* Clinically significant diseases or abnormal laboratory values as assessed during the screening medical history, physical exam, and laboratory evaluations.
* A history (within the past year) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurologic disease. The exclusion criteria also includes 1) positive urine pregnancy test 2) The use of oral contraceptives 3) The lack of use of acceptable barrier methods of birth control unless abstinent
* Use of any concomitant medication including herbal medications or a history of hypersensitivity to the medications used in the study
* History of sensitivity to CB juice or products
* Poor metabolizers of CYP2D6
* Active smoking or use of caffeine-containing beverages for 2 weeks prior to and during the study
* Inability to conform with dietary restrictions required for the study
* Drug or alcohol abuse (more than 3 drinks/day)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Donovan, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States